CLINICAL TRIAL: NCT01666834
Title: Southeast Univerity
Brief Title: Cross-section Survey of Mechanical Ventilation and Acute Respiratory Distress Syndrome in China
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Ling Liu, Dr., Southeast University, China
Other Study IDs: zdyyicu3
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2013-05

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: mechanical ventilation, ARDS, Ventilator strategy, outcome
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The characteristics and outcomes of a mixed group of critically ill patients who received mechanical ventilation are not known in China.

A 1 month Cross-section survey will be performed with the aim of describing the characteristics and outcomes of conventional mechanical ventilation and treatment of acute respiratory distress syndrome in intensive care units in China.

DETAILED DESCRIPTION:
From August 31th 2012 to September 30th 2012, all patients admit to ICUs were screened, mechanical patients and patients with ARDS be enrolled. The demographic characteristics, diagnosis, formerly medical history, Ventilator indications, Ventilator data, other respiratory treatments, weaning outcome and 28 day mortality, and the treatment of ARDS will be recorded.

ELIGIBILITY:
Inclusion Criteria for mechanical ventillation patients:

Meet one of the following criteria

1. Patients who were admitted to ICU from September 1st to 31th 2012, and received invasive mechanical ventilation for more than 24 hours
2. Patients who were admitted to ICU from September 1st to 31th 2012, and received non-invasive mechanical ventilation for more than 12 hours
3. Patients who were admitted to ICU from September 1st to 31th 2012, and who fulifll the ARDS Berlin Definition or AECC Definiton

Exclusion Criteria:

1. lesson than 18 years old or more than 85 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A mixed group of critically ill patients who received mechanical ventilation or patient with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
percentange of mechanical ventilation | 1 month
  in the onw month period, How many patients in the intensive care unit are ventilated.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, professor, Study Director — southeast university
Locations (1):
- Zhong-Da hospital, southeast univerty, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xie J, Liu L, Yang Y, Yu W, Li M, Yu K, Zheng R, Yan J, Wang X, Cai G, Li J, Gu Q, Zhao H, Mu X, Ma X, Qiu H. A modified acute respiratory distress syndrome prediction score: a multicenter cohort study in China. J Thorac Dis. 2018 Oct;10(10):5764-5773. doi: 10.21037/jtd.2018.09.117. PMID 30505484
- [Derived] Liu L, Yang Y, Gao Z, Li M, Mu X, Ma X, Li G, Sun W, Wang X, Gu Q, Zheng R, Zhao H, Ao D, Yu W, Wang Y, Chen K, Yan J, Li J, Cai G, Wang Y, Wang H, Kang Y, Slutsky AS, Liu S, Xie J, Qiu H. Practice of diagnosis and management of acute respiratory distress syndrome in mainland China: a cross-sectional study. J Thorac Dis. 2018 Sep;10(9):5394-5404. doi: 10.21037/jtd.2018.08.137. PMID 30416787